CLINICAL TRIAL: NCT03566212
Title: Clinical Comparative Study of Efficacy of Camouflaged Syringe vs Conventional Syringe in Reducing Dental Anxiety
Brief Title: Efficacy of Camouflaged Syringe vs Conventional Syringe
Acronym: ECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sneha D. Suwarnkar (Other)
Responsible Party: Sponsor-Investigator, Sneha D. Suwarnkar, Principal investigator, Saraswati-Dhanwantari Dental College & Hospital
Organization: Saraswati-Dhanwantari Dental College & Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaraswatiDhanwantari
Record Dates: First submitted 2018-05-30; First posted 2018-06-25 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Dental Anxiety; Behavior
Keywords: Anxiety; Camouflaged syringe; Conventional syringe
MeSH Terms: conditions — Behavior; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: local anesthesia is administered by using either camouflaged syringe or conventional syringe and was compared for reduction in anxiety levels in both groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional syringe (Experimental): Individuals requiring local anesthesia for dental treatment were treated in first group by using conventional syringe.
  Interventions: Device: Conventional Syringe
- camouflaged syringe (Experimental): Individuals requiring local anesthesia for dental treatment were treated in second group by using camouflage syringe.
  Interventions: Device: Camouflage Syringe

INTERVENTIONS:
Device: Conventional Syringe — local anesthesia was administered in first group using Conventional syringe
  Arms: conventional syringe
Device: Camouflage Syringe — local anesthesia was administered in second group using Camouflage syringe
  Arms: camouflaged syringe

SUMMARY:
This study evaluates the efficacy of Camouflage syringe vs Conventional syringe in reducing Dental Anxiety and increasing behaviour rating.Half of the participants received local anesthesia using camouflaged syringe, while others received using conventional syringe.

DETAILED DESCRIPTION:
Dental anxiety and phobia result in avoidance of dental care. Since the injection itself can be painful, pain reduction procedures warrant continued investigation. Camouflage design deals with the visual impact of the needle and syringe though the tactile sensation remains unaltered. In our study, post treatment anxiety levels in camouflaged syringe was reduced as compared to conventional syringe group and this might be because, patients with low anxiety tend to have high pain thresholds.

ELIGIBILITY:
Inclusion Criteria:

* retained teeth,
* badly carious teeth,
* mobile teeth
* requiring a dental procedure under local anesthesia were selected.

Exclusion Criteria:

* Mentally challenged children
* those with medical conditions contraindicating the use of local anesthesia and / or surgical procedures

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-08-13 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Anxiety levels by using the Chotta Bheem and Chutki scale | after 5 minutes
  Anxiety levels in both camouflaged group and conventional group in the children were scored before and after the procedure using the Chotta Bheem and Chutki scale. The Chotta Bheem and Chutki (CBC) scale comprises two separate cards: one for boys and the other for girls. The cartoon characters of Chotta Bheem and Chutki were chosen to depict various emotions for boys and girls respectively. Each card consists of a series of six figures depicting sequentially various emotions from 'happy' to 'unhappy and running away' of the cartoon character. Score 1 is happy face, score 2 is sad face, score 3 is crying face, score 4 is angry face, score 5 is shouting and score 6 is running. So, here, score 1 depicts patient is happy whereas as score increases anxiety level also increases which denotes that patient is unhappy.

SECONDARY OUTCOMES:
Behavior rating by using Frankel Behaviour rating scale | after 10 minutes
  Behavior rating in both camouflaged group and conventional group in the children were scored before and after the procedure using Frankel Behaviour rating scale. Behavior rating scale comprised of scores from definitely negative to definitely positive. 'Double negative'(--) i.e. 'definitely negative' score indicates that patient refuses treatment, 'negative score'(-) indicates that patient is reluctant to accept treatment, there is evidence of negative attitude but not pronounced, ' positive score' (+) indicates that patient accepts treatment though there is cautious with treatment but follows dentist's instructions cooperatively whereas ' definitely positive score' (++) indicates that there is good raport of patient with dentist and accepts the treatment with enjoyment. So, as score increases from definitely negative to definitely positive, behaviour of children also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Sneha D Suwarnkar, MDS, Principal Investigator — Saraswati Dhanwantari Dental College and Hospital, Parbhani
Locations (1):
- Dr Sneha D Suwarnkar, Parbhani, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
it will be dependent on publication